CLINICAL TRIAL: NCT04775329
Title: Primary Prophylaxis for Spontaneous Bacterial Peritonitis in Decompensated Chronic Liver Disease With Small Bowel Bacterial Overgrowth: A Randomised Trial
Brief Title: Primary Prophylaxis for Spontaneous Bacterial Peritonitis
Acronym: SIBOC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow recruitment and study closure
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SIBOC
Record Dates: First submitted 2021-01-25; First posted 2021-03-01 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Decompensated Cirrhosis; Small Bowel Bacterial Overgrowth Syndrome
Keywords: Rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomised, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Standard of care
- Treatment arm (Active Comparator)
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 1000mg OM
  Arms: Treatment arm

SUMMARY:
Patient with liver cirrhosis commonly have co-existing small bowel bacterial overgrowth (SIBO) yet may be asymptomatic. It is unclear as to the value of treating SIBO in asymptomatic individuals. Cirrhosis increase permeability of the gastrointestinal mucosa. It is postulated that in cirrhosis, endotoxins translocate across the gut mucosal barrier resulting in a second hit within hepatocyte perpetuating decompensation and spontaneous bacterial peritonitis. We hypothesise that cirrhosis patients with concomitant SIBO are particularly vulnerable for endotoxin translocation and would benefit from treatment. Treatment of SIBO would reduce the risk of spontaneous bacterial peritonitis and other liver-related morbidities. We aim to treat a cohort of patients with severe liver disease and concomitant SIBO with antibiotics as prophylaxis and compare the risk of spontaneous bacterial peritonitis, further liver-related morbidity and survival against untreated asymptomatic controls.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated liver cirrhosis (Childs B & C) with ascites.
* Established diagnosis of SIBO

Exclusion Criteria:

* Known allergy to treatment drugs
* Inability to undergo test confirm the success of SIBO eradication;
* Pregnant or lactating women
* Terminal malignancy.
* Untreated Viral Hepatitis
* Alcoholic Liver disease with ongoing drinking.
* Respiratory Failure
* Recent antibiotics and proton-pump inhibitor within 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Spontaneous bacterial peritonitis | 12 months
  To determine the rate of cirrhosis-related complications, with and without Rifaximin among decompensated cirrhosis with SIBO.

SECONDARY OUTCOMES:
Incidence of all liver related events (hepatic encephalopathy, variceal bleeding, acute on chronic liver failure) | 12 months
  To study and understand the immunophysiological and gut microbiota changes associated with bowel decontamination among cirrhosis patients with SIBO using serum biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: YU JUN WONG, MD, MRCP FAMS, Principal Investigator — Changi General Hospital
Locations (1):
- Wong Yu Jun, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180